CLINICAL TRIAL: NCT01850485
Title: Microcirculatory Perfusion as Measured by Sublingual SDF Imaging and NIRS in Patients With Coma After Out-of-hospital Cardiac Arrest Treated With Mild Therapeutic Hypothermia (TH) or Not Treated With Mild-TH
Brief Title: Microcirculatory Perfusion in Patients With Coma After Out-of-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, RN, Frisius Medisch Centrum
Other Study IDs: TPO 745
Record Dates: First submitted 2012-04-23; First posted 2013-05-09 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; therapeutic hypothermia; microcirculation
MeSH Terms: conditions — Heart Arrest | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normothermia, 36 degrees: microcirculation after cardiac arrest by SDF and NIRS, in patients treated with 36 degrees, difference is temperature, in this group 36
  Interventions: Device: microcirculation by SDF and NIRS, in 33 and 36 degrees
- 33 degrees, therapeutic hypothermia: microcirculation after cardiac arrest by SDF and NIRS, in patients treated with 33 degrees, difference is temperature, in this group 33
  Interventions: Device: microcirculation by SDF and NIRS, in 33 and 36 degrees

INTERVENTIONS:
Device: microcirculation by SDF and NIRS, in 33 and 36 degrees — at baseline, after 12 and 24 hours in both arms
  Other Names: measurements of the microcirculation by SDF and NIRS; in both arms

SUMMARY:
The hypothesis is: In patients after an out of hospital cardiac arrest, treated with therapeutic hypothermia (33°C) will be found significantly more microcirculatory abnormalities, compared to the same group of patients treated with 36°C.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the (sublingual) microcirculation in patients after an out of hospital cardiac arrest (OHCA). The microcirculation is measured in this study by Sublingual Side Stream Darkfield (SDF) Imaging and Near InfraRed Spectroscopy (NIRS) at admission and after 12 and 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest
* > 18 years
* informed consent
* ROSC (return of spontaneous circulation) < 4 hours

Exclusion Criteria:

* recent maxillofacial surgery
* participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients after out of hospital cardiac arrest
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matty Koopmans, RN, Principal Investigator — medical center leeuwarden
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Netherlands

REFERENCES:
- [Derived] Koopmans M, Kuiper MA, Endeman H, Veenstra G, Vellinga NA, de Vos R, Boerma EC. Microcirculatory perfusion and vascular reactivity are altered in post cardiac arrest patients, irrespective of target temperature management to 33 degrees C vs 36 degrees C. Resuscitation. 2015 Jan;86:14-8. doi: 10.1016/j.resuscitation.2014.09.025. Epub 2014 Oct 18. PMID 25449350

RESULTS

PARTICIPANT FLOW:
Groups:
- Normothermia, 36 Degrees: microcirculation after cardiac arrest by SDF and NIRS, in patients treated with 36 degrees
  microcirculation by SDF and NIRS, in 33 and 36 degrees: at baseline, after 12 and 24 hours in both arms
- 33 Degrees, Therapeutic Hypothermia: microcirculation after cardiac arrest by SDF and NIRS, in patients treated with 33 degrees
  microcirculation by SDF and NIRS, in 33 and 36 degrees: at baseline, after 12 and 24 hours in both arms
Period: Overall Study
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia
Started | 9 | 13
Completed | 9 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia | Total
Number analyzed (Participants) | 9 | 13 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (12.4) | 68.9 (9.3) | 66.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 6 | 12 | 18
Region of Enrollment [Number; unit: participants]
  Netherlands | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Microvascular Flow Index (MFI)
Description: Microvascular Flow Index; minimum score = 0 (= no flow) and maximum score = 3 (=normal flow)
Time Frame: baseline measurement
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia
Number analyzed (Participants) | 9 | 13
units on a scale | 1.7 [0.7 to 2.4] | 1.1 [0.4 to 1.9]

2. Secondary Outcome: RincStO2
Description: tissue oxygenation measured by Near Infrared Spectroscopy
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia
Number analyzed (Participants) | 9 | 13
percent saturation | 44.6 (15.8) | 58.9 (13.5)

3. Secondary Outcome: Fluid Balance After 24 Hours
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia
Number analyzed (Participants) | 9 | 13
liters | 1.79 (0.92) | 3.33 (1.18)

4. Secondary Outcome: Inotropes and Vasopressor Dose
Time Frame: baseline
Measure: Median (Inter-Quartile Range); unit: mcg/kg/min
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia
Number analyzed (Participants) | 9 | 13
mcg/kg/min | 0.00 [0.00 to 1.9] | 0.00 [0.00 to 4.89]

5. Secondary Outcome: Cardiac Index
Description: Cardiac Index is cardiac output indexed for body weight
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: L/m2
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia
Number analyzed (Participants) | 9 | 13
L/m2 | 2.1 (0.64) | 1.9 (0.73)

6. Secondary Outcome: Lactate
Description: lactate levels in serum
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia
Number analyzed (Participants) | 9 | 13
mmol/l | 1.71 (0.48) | 2.78 (1.1)

7. Secondary Outcome: SvO2
Description: (venous oxygen saturation)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia
Number analyzed (Participants) | 9 | 13
percent saturation | 61.2 (13.6) | 69.4 (10.3)

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Normothermia, 36 Degrees | 33 Degrees, Therapeutic Hypothermia
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 0/9 | 0/13

LIMITATIONS AND CAVEATS:
Relative small sample size Large inter individual variability in microvascular reactivity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes